CLINICAL TRIAL: NCT07315490
Title: A Comparison of the Effect of Air Versus Lignocaine for Endotracheal Tube Cuff Inflation on Postoperative Sore Throat and Intracuff Pressure
Brief Title: Air Versus Lignocaine for Endotracheal Tube Cuff Inflation and Effect on Postoperative Sore Throat and Intracuff Pressure
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PAEC General Hospital, Islamabad (Other)
Responsible Party: Principal Investigator, Zubaria Liaquat, Post Graduate Trainee, Department of Anesthesiology, PAEC general hospital Islamabad, PAEC General Hospital, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PGHI-IRB (DMe)-RCD-06-096
Record Dates: First submitted 2025-12-05; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Sore Throat, Cough, Hoarseness
Keywords: Endotacheal Tube; General Anesthesia; Air; ETT cuff; Xylocaine; Post operative sore throat; ETT cuff Manometer; Cough; Sore throat; Hoarseness of voice; Intra cuff pressure
MeSH Terms: conditions — Cough; Hoarseness; Pharyngitis | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylocaine (Experimental): In 50% of subjects undergoing surgeriws under GA, Xylocaine will be used for ETT cuff inflation. Intracuff pressures will be measured every 15 mins using ETT cuff manometer and compared with intracuff air.Postoperative POST scoring will be done to study its effect on postopertaive sorethroat and incidence will weighed against intracuff air.
  Interventions: Drug: Xylocaine
- Air (Placebo Comparator): In 50% of subjects undergoing surgeries under GA, air will be ussed for ETT cuff inflation, intracuff pressures will be measured every 15 min POST scoring will be done postoperatively.
  Interventions: Drug: Xylocaine

INTERVENTIONS:
Drug: Xylocaine — In patients undergoing surgeries under GA, xylocaine will be used for 50% subjects and ETT cuff pressures will be measured at regular and compated to air to study if using xylocaine can abolish the affect of Nitrous oxide on intracuff air pressure. Also postoperatively, POST scoring will be done.

SUMMARY:
Endotracheal Tube (ETT) is frequently used for GA (general anesthesia) to deliver oxygen and volatile anesthetic agents to the patient and serves as a channel for anesthetic gases. The ETT cuff helps in positive pressure ventilation and maintains an adequate seal between the endotracheal tube and trachea.

Prolonged inflation of ETT cuff can cause ischemic changes of tracheal mucosa and other complications like postoperative sore throat (POST), hoarseness of voice, difficulty in swallowing, tracheal wall ulcer, stricture etc. Among these, the occurrence of sore throat after GA ranges from 21 - 65% Hence it important to measure ETT cuff pressure in intubated patients. The reliable and convenient way for this is using an ETT manometer, which is not readily available in most of hospitals in Pakistan.Many studies have focused on incidence of POST. Most of these studies have been done in western population and differences in various ethnicities are well reported . In Pakistan, air is widely used for ETT cuff inflation.

If the results depict minimal cuff pressure changes and postoperative side effects with Xylocaine as compared to air, then it can be inferred that cuff pressure does not increase due to N2O when Xylocaine is used, hence, it can be safely used for cuff inflation eliminating the requirement of ETT cuff pressure monitoring and also the ETT cuff manometer, serving as a cost-effective alternative.

DETAILED DESCRIPTION:
Every patient will be evaluated in the preoperative clinic where detailed present and past history including any current illness, medication, previous surgeries and addiction will be taken and recorded. Also baseline investigations will be evaluated. Airway examination and Mallampati scoring will be done. The patients will be divided into 2 groups: Group A (Air) and Group X (Xylocaine plain 2%), using air and Xylocaine for alternate patients.

In the OT, an anesthesia resident will record baseline vitals. An IV line with 18 or 20 G cannula will be secured and IV fluid Ringer Lactate will be infused according to the body weight. All patients will be preoxygenated for 3min. Patients will be premedicated Ondansetron 0.8mg/kg, Glycopyrrolate 0.2mg/kg, Dexamethasone 8mg, inducted with Propofol 2mg/kg, Atracurium 0.5mg/kg. Anesthesia will be maintained with Oxygen 50%, Nitrous oxide 50% and Isoflurane. Patient will be intubated with a cuffed ETT, size 7 or 7.5 mm for males and 6.5 or 7mm for females. For Group A the cuff of the ETT will be inflated with air and for Group X the ETT cuff will be inflated with Xylocaine plain 2% and the ETT cuff pressure will be measured by an anesthesia assistant using cuff manometer immediately after intubation and at 5, 15, 30min and then at every 30 min till the completion of surgery.

On completion of surgery, anesthesia will be reversed by weaning of the anesthetic gases and neostigmine 0.05-0.07mg/kg with glycopyrrolate will be used to reverse the remaining muscle paralysis. When the patient is awake the ETT cuff will be deflated by removing the inflating agent. Then the patient will be oxygenated with a face mask until needed. Signs and symptoms like postoperative sore throat, cough and hoarseness of voice will be recorded immediately after extubation and at 30min, 6hr and 24 hr post operatively. The severity of POST will be scored on a scale of 0-3 (0: No POST; 1: Mild; 2: Moderate; 3: Severe).

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anaesthesiologists) I and II
* Male/Female
* Age group 18 - 55 years
* Patient undergoing surgery under general anesthesia.
* Patients undergoing surgery in supine/ Trendelenburg position.

Exclusion Criteria:

* ASA III and IV
* Patients with preoperative history of cough or sore throat
* Patients undergoing nose, throat, or airway surgery.
* Patients with history of allergic diseases
* Patient with known pulmonary disease
* Patients in whom more than 1 attempt on intubation is done
* Patients who may need postoperative ventilation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-02 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of ETT cuff Pressure | From the time of intubation till extubation
  Patients will be divided in 2 groups on basis of the medium used for ETT cuff infalation (Air or Xylocaine) and intracuff pressure will be measured using ETT cuff manometer immediately after intubation, at 5min, 15min, 30min and then eveey 30 min till completion of surgery
Postoperative Sorethroat, Cough and Hoarseness | From extubation till 24 hours postoperatively
  This will be measured immediately after extubation, at 30min, 6hrs and 24 hours postoperative using POST (postoperative sorethroat) scoring scale for both groups of subjects and responses will be compared.
  Sorethroat (grade 0-3; where 0 stand for no sorethroat and 3 stand for severe sorethroat) Cough (grade 0-3; where 0 stand for no cough and 3 stand for severe cough) Hoarseness of Voice (grade 0-3; where 0 stand for no hoarseness and 3 stand for severe hoarseness)

SECONDARY OUTCOMES:
Demographic data | From enrollment till 24 hours postoperatively
  Age: can affect airway anatomy (loss of elasticity, missing or loose teeth) BMI: higher malampatti scores, difficult intubation (kg/m²) Gender: structural airway differences, different ETT sizes Difficulty of intubation: directly related to airway trauma Duration of surgery: directly related to increase in cuff pressures in N2O anesthesia (in minutes) ASA physical status: according to classification given by Amercian Society of Anesthesiologists, will be done preoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat, Islamabad, Federal Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Changes in endotracheal tube cuff pressures and incidence of post-operative sore throat while using different inflating agents — https://doi.org/10.3329/jbcps.v42i1.70624
- See also: Postoperative Sore Throat Following General Surgical Procedures under General Anesthesia with Endotracheal Intubation — https://orcid.org/0009-0004-4811-1903
- See also: Effect of Air versus 1% Lignocaine used for Endotracheal Tube Cuff Inflation on Laryngotracheal Morbidity after Laparoscopic Surgery- A Randomised Clinical Study — https://www.jcdr.net/articles/PDF/17097/57885_CE(AD)_F(SHU)_PF1(SC_SHU)_PFA(SS)_PB(SC_SS)_PN(SS).pdf